CLINICAL TRIAL: NCT04480307
Title: A Randomized, Double-Blind, Placebo Controlled Trial, Examining the Safety, Tolerability, Pharmacodynamic Effects and Pharmacokinetics of Temelimab Following Rituximab Treatment in Patients With Relapsing Forms of Multiple Sclerosis (RMS)
Brief Title: Clinical Trial Assessing Temelimab Following Rituximab Treatment in Patients With Relapsing Forms of Multiple Sclerosis
Acronym: ProTEct-MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GeNeuro Innovation SAS (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-401; 2019-004822-15 (EudraCT Number)
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Forms of Multiple Sclerosis; GNbAC1; Human Endogenous Retrovirus Type W; HERV-W; Temelimab
MeSH Terms: conditions — Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- temelimab 18 mg/kg (Experimental): Monthly IV repeated dose
  Interventions: Drug: temelimab 18 mg/kg
- temelimab 36 mg/kg (Experimental): Monthly IV repeated dose
  Interventions: Drug: temelimab 36 mg/kg
- temelimab 54 mg/kg (Experimental): Monthly IV repeated dose
  Interventions: Drug: temelimab 54 mg/kg
- Placebo (Placebo Comparator): Monthly IV repeated dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: temelimab 18 mg/kg — temelimab 18 mg/kg will be given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
  Arms: temelimab 18 mg/kg
Drug: temelimab 36 mg/kg — temelimab 36 mg/kg will be given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
  Arms: temelimab 36 mg/kg
Drug: temelimab 54 mg/kg — temelimab 54 mg/kg will be given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
  Arms: temelimab 54 mg/kg
Drug: Placebo — Placebo will be given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled Phase IIa clinical study, assessing safety, tolerability, pharmacodynamic effects and pharmacokinetics of temelimab, administered at three different dose levels (18 mg/kg or 36 mg/kg or 54 mg/kg).

In this study temelimab is administered subsequently to rituximab therapy, i.e. no co-administration of rituximab and temelimab is done in this study.

ELIGIBILITY:
Main Inclusion Criteria:

* Current diagnosis of RMS, based on McDonald 2017 criteria
* Having received treatment with rituximab, as per local clinical routine for at least 12 months prior to the Screening Visit
* Having received their last dose of rituximab not more than 8 weeks and not less than 4 weeks before Randomization (Study Day 1)
* Having expanded disability status scale (EDSS) 2.5 - 5.5 inclusive at Screening
* Present clinical worsening in one or more neurological domains as assessed by EDSS, ambulatory function as assessed by 6MWT or T25FW, cognitive functioning as assessed by SDMT or increased need of walking aids or pharmacological/procedures for bowel and bladder functions over the last year.

Main Exclusion Criteria:

* Current diagnosis of primary progressive MS (PPMS)
* Any disease other than MS (e.g. myelitis and /or bilateral optic neuritis) that could better explain the patient's signs and symptoms
* Usage of any of the following medications prior to the Screening visit:

  * Any usage of interferon beta, glatiramer acetate, IV immunoglobulin (IVIG), dimethyl fumarate or teriflunomide within 12 months prior to Screening,
  * Any history of exposure to mitoxantrone, cladribine, alemtuzumab, cyclophosphamide, systemic cytotoxic therapy, total lymphoid irradiation, and/or bone marrow transplantation at any time,
  * Any usage of natalizumab within 24 months prior to Screening,
  * Any usage of highly potent immune modulating therapy, such as: ocrelizumab, ofatumumab, fingolimod, siponimod, ozanimod or anti-cytokine therapy, plasmapheresis or azathioprine within 12 months prior to Screening,
  * Any usage of any experimental treatment if not washed out for ≥ 5 half-lives or ≥ 12 months (whichever is longer), except rituximab which is allowed before the study.
* CTCAE Grade 2 or greater lymphopenia
* Any major medical or psychiatric disorder that would affect the capacity of the patient to fulfill the requirements of the study
* History or presence of serious or acute heart disease such as uncontrolled cardiac dysrhythmia or arrhythmia, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure (NYHA class 3 or 4)
* Any history of cancer with the exceptions of basal cell carcinoma and/or carcinoma in situ of the cervix, and only if successfully treated by complete surgical resection, with documented clean margins and any medically unstable condition as determined by the investigator
* Pregnant or breastfeeding women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Leppert, MD, Study Director — GeNeuro Innovation SAS
Locations (1):
- Center for Neurology, Academic Specialist Center, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening details:
  Subjects who met the inclusion criteria at the Screening visit (within 3 weeks prior to dosing) and at the Baseline visit (Study Day 1 (SD1)) were considered eligible to participate in the clinical study.
Groups:
- Temelimab 18 mg/kg: Temelimab 18 mg/kg was given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
- Temelimab 36 mg/kg: Temelimab 36 mg/kg was given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
- Temelimab 54 mg/kg: Temelimab 54 mg/kg was given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
- Placebo: Placebo was given as monthly (4-weekly) intravenous (IV) infusions over 48 weeks (12 administrations in total).
Period: Overall Study
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
Started | 11 | 10 | 10 | 10
Completed | 11 | 9 | 10 | 9
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomised set (RS): All patients to whom a therapeutic treatment was randomly assigned using an interactive response system. Patients were analysed in their randomisation group whatever the treatment they received
Groups:
- Total: Total of all reporting groups
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 10 | 10 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (7.3) | 47.9 (6.3) | 45.2 (10.2) | 45.6 (9.4) | 45.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 3 | 6 | 21
  Male | 4 | 5 | 7 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 9 | 10 | 39
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Sweden | 11 | 10 | 10 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Analysis of Adverse Events (AEs) focused on Treatment Emergent AEs (TEAEs)
Time Frame: 48 weeks
Population: Safety set (SAF): all patients having taken at least one dose of IMP. Patients were allocated to the group based on treatment they received
Measure: Number; unit: Participants with at least one TEAE
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
Number analyzed (Participants) | 11 | 10 | 10 | 10
Participants with at least one TEAE | 10 | 9 | 10 | 9

2. Secondary Outcome: Neuroimaging
Description: Change in magnetization transfer saturation (MT Sat) in periventricular NAWM at Week 48 compared to Baseline. The MT Sat represents the fraction of free water, as transformed to per-unit scale, saturated by a single Magnetization transfer (MT) pulse during repetition time (TR).
Time Frame: 48 weeks
Population: Per protocol (PP) set: All patients of the RS with no major protocol deviations and with at least 9 infusions performed. All protocol deviations were assessed and documented on a case-by-case basis prior to database lock, and deviations considered to have a serious impact on the efficacy results led to the relevant patient being excluded from the set.
Measure: Mean (Standard Deviation); unit: per unit
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
Number analyzed (Participants) | 9 | 9 | 7 | 8
per unit | -0.011 (0.097) | -0.060 (0.081) | -0.016 (0.194) | 0.008 (0.113)
Statistical Analysis 1: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; Test type: Superiority; p = 0.5084, ANCOVA; LS Mean Difference = -0.031, 95% CI 2-sided [-0.124 to 0.063]
Statistical Analysis 2: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; Bayesian analysis is done using a non-informative prior on the mean observed difference; Test type: Superiority; Bayesian; Difference of change from baseline a posteriori; Difference of change from Baseline = -0.021, 95% CI 2-sided [-0.121 to 0.057]

3. Secondary Outcome: Neuroimaging
Description: Change in magnetization transfer saturation (MT Sat) in cortex at Week 48 compared to Baseline. The MT Sat represents the fraction of free water, as transformed to per-unit scale, saturated by a single Magnetization transfer pulse during repetition time.
Time Frame: 48 weeks
Population: PP set
Measure: Mean (Standard Deviation); unit: per unit
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
Number analyzed (Participants) | 9 | 9 | 6 | 7
per unit | 0.037 (0.058) | 0.044 (0.044) | -0.013 (0.077) | 0.018 (0.040)
Statistical Analysis 1: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; Test type: Superiority; p = 0.9472, ANCOVA; LS Mean Difference = -0.002, 95% CI 2-sided [-0.052 to 0.049]
Statistical Analysis 2: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; Bayesian analysis is done using a non-informative prior on the mean observed difference; Test type: Superiority; Bayesian; Difference of change from Baseline a posteriori; Difference of change from Baseline = 0.012, 95% CI 2-sided [-0.036 to 0.059]

4. Secondary Outcome: Neuroimaging
Description: Change in T1 and T2 lesion volume at Week 48 compared to Baseline
Time Frame: 48 weeks
Population: PP set
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 8
mL
  Change in T1 lesion volume | -0.055 (0.315) | -0.032 (0.686) | 0.227 (0.405) | -0.044 (0.185)
  Change in T2 lesion volume | 0.028 (0.085) | 0.029 (0.088) | 0.023 (0.061) | 0.027 (0.075)
Statistical Analysis 1: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; ANCOVA analysis for T1 lesion volume parameter; Test type: Superiority; p = 0.4027, ANCOVA; LS Mean Difference = 0.154, 95% CI 2-sided [-0.216 to 0.524]
Statistical Analysis 2: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; ANCOVA analysis for T2 lesion volume parameter; Test type: Superiority; p = 0.7428, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.051 to 0.071]

5. Secondary Outcome: Neuroimaging
Description: Change in brain parenchymal volume fraction at Week 48 compared to Baseline. The brain parenchymal fraction is defined as the ratio of brain parenchymal volume to the total volume within the brain surface contour.
Time Frame: 48 weeks
Population: Per protocol (PP) set
Measure: Median (Standard Deviation); unit: Ratio
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 8
Ratio | -0.013 (0.011) | -0.021 (0.032) | -0.011 (0.013) | -0.019 (0.017)
Statistical Analysis 1: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; Test type: Superiority; p = 0.7314, ANCOVA; LS Mean Difference = 0.003, 95% CI 2-sided [-0.013 to 0.018]
Statistical Analysis 2: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; Bayesian analysis is done using a non-informative prior on the mean observed difference; Test type: Superiority; Bayesian; Difference of change from Baseline a posteriori; Difference of change from Baseline = 0.005, 95% CI 2-sided [-0.010 to 0.023]

6. Secondary Outcome: Neuroimaging
Description: Change in thalamic volume fraction at Week 48 compared to Baseline. The thalamic volume fraction is the ratio of the legitimate (i.e. thalamic) brain tissue volume to the total volume within the brain surface contour.
Time Frame: 48 weeks
Population: PP set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 8
Ratio | -0.000 (0.000) | -0.000 (0.000) | -0.000 (0.000) | -0.000 (0.000)
Statistical Analysis 1: Comparison: Temelimab 18 mg/kg vs Temelimab 36 mg/kg vs Temelimab 54 mg/kg; Test type: Superiority; p = 0.7662, ANCOVA; LS Mean Difference = 0, 95% CI 2-sided [0 to 0]

ADVERSE EVENTS:
Time Frame: The collection of Adverse Events (AEs) was from the time the patient signed the informed consent onwards up to Week 48.
Description: Analysis of Adverse Events (AEs) focused on Treatment Emergent AEs (TEAEs).
Arm/Group | Temelimab 18 mg/kg | Temelimab 36 mg/kg | Temelimab 54 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/11 | 9/10 | 10/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temelimab 18 mg/kg (N=11) | Temelimab 36 mg/kg (N=10) | Temelimab 54 mg/kg (N=10) | Placebo (N=10)
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temelimab 18 mg/kg (N=11) | Temelimab 36 mg/kg (N=10) | Temelimab 54 mg/kg (N=10) | Placebo (N=10)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 5 (5) | 3 (3)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04480307/Prot_SAP_000.pdf